CLINICAL TRIAL: NCT06968169
Title: The Short-term Verbal Memory Endophenotype for Developmental Language Disorder
Brief Title: The Short-term Verbal Memory Endophenotype for Developmental Language Disorder Language Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Father Flanagan's Boys' Home (Other)
Collaborators: University of Iowa (Other); National Institutes of Health (NIH) (NIH); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 24-18-XP; R01DC011742 (NIH)
Record Dates: First submitted 2025-02-24; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Developmental Language Disorder; Healthy Subjects
Keywords: nonword repetition; word learning; memory; attention
MeSH Terms: conditions — Language Development Disorders | interventions — MAP Kinase Signaling System

STUDY DESIGN:
Intervention Model Description: Aims 1 and 2 are single group interventions. Aim 3 is not an intervention. Aim 4 is a parallel intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Prosody (Experimental): In Aim 1a, the syllables to be repeated are presented with English-like prosody or list-like prosody.
  Interventions: Behavioral: Supportive learning
- Meaning (Experimental): In Aim 1a, the syllables to be repeated will have meaning (e.g., neck) or no meaning (e.g., ba).
  Interventions: Behavioral: Supportive learning
- Grammar (Experimental): In Aim 1b, the syllables to be repeated are English adjectives and nouns. They will be presented to obey English grammar (e.g., happy pencil) or not (e.g., pencil happy).
  Interventions: Behavioral: Supportive learning
- Attention (Experimental): In Aim 2, the syllables to be repeated will be presented in the 'baseline' condition or an 'attention-grabbing' condition. The attention grabbers are a reduction in the audio signal of 10dB (so that the child must listen carefully) and a visual cue (a cartoon character with large ears to cue listening carefully).
  Interventions: Behavioral: Supportive learning
- Encoding (Experimental): In Aim 4, new words will be learned from instruction that involves active practice (high encoding condition) or passive study (low encoding condition).
  Interventions: Behavioral: Cascades

INTERVENTIONS:
Behavioral: Supportive learning — All interventions are manipulations to the stimuli that the child hears with the goal of discovering which manipulations support verbal learning.
  Arms: Attention; Grammar; Meaning; Prosody
Behavioral: Cascades — The intervention is a manipulation of word instruction with the goal of discovering whether weaker word learning results in cascading effects on semantic category memory and sentence comprehension.
  Arms: Encoding

SUMMARY:
The goal of this clinical trial is to determine how memory and attention affect the ability of children with developmental language disorder (DLD) to learn and use new vocabulary.

DETAILED DESCRIPTION:
The goal of this clinical trial is to determine how memory and attention affect the ability of children with developmental language disorder (DLD) to learn and use new vocabulary.

Aims 1-3 include children with DLD and healthy children with typical language development. The general hypothesis is that the memory and attention challenges that characterize DLD, but not healthy development, affect the robustness of word learning. Aim 4 includes healthy children only to simulate the cascading effects of weak word learning on the broader linguistic system. The main questions this clinical trial aims to answer are:

What is the role of linguistic long-term memory in children's ability to hold new verbal information in short-term memory? What is the role of attention in children 's ability to hold new verbal information in short-term memory? What are the cascading effects of short-term verbal memory problems on the integrity of the language system?

In Aim 1a, researchers will compare syllable repetitions when those syllables do or do not have English-like prosody and do or do not have meaning to see if knowledge of prosody and word meaning supports accurate short-term memory.

In Aim 1b, researchers will compare the repetition of adjectives and nouns when those words do or do not have English-like grammar (i.e., when they are presented as adjective + noun rather than noun + adjective) to see if knowledge of word order supports accurate short-term memory.

In Aim 2, researchers will compare the syllable repetitions when those syllables are presented with or without attention cues and with or without a delay of 500msec between presentation and response to see if attention facilitates accurate short-term memory. The delay condition is intended to increase load on short-term memory.

In Aim 3, all measures are observational. The researchers will assess the child's long-term memory of language, attention skills, and verbal short-term memory to see if children with DLD but good attention skills are able to perform well on short-term memory tasks.

In Aim 4, researchers will compare the ability of children to comprehend newly learned words that are taught via active retrieval or passive study. Active retrieval yields more robust learning, and passive study yields weaker learning. The goal is to compare how well children use those newly learned words to recall semantic category information (e.g., was it a bug or a bird) and comprehend sentences to see if the weak word learning has cascading impacts beyond learning the word itself.

ELIGIBILITY:
Inclusion Criteria:

* Has DLD or typical language development

Exclusion Criteria

* Has not been exposed to English since birth
* Has other neurodevelopmental or sensory condition that could explain the language problem (e.g., intellectual disability, autism, hearing loss).

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-02-09 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Syllable Repetition | Day 1
  Number of syllables pronounced correctly.
Accuracy of Word Comprehension | Day 2
  Number of correct answers on a 4-alternative-forced-choice word comprehension probe.

CONTACTS AND LOCATIONS:
Overall Officials: Karla McGregor, Ph.D., Principal Investigator — Boystown National Research Hospital
Locations (1):
- Boys Town National Research Hospital, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
The study team will share research data generated and metadata and descriptors. The purpose is to make shared data meaningful and usable by other researchers. The data will be behavioral data generated from clinical measures and behavioral experiments. The data will consist of numbers (e.g., accuracy levels, scores), demographic descriptors (e.g., age and sex), and audio files of children's repetitions of word- and nonword syllables. De-identified, individual-level raw data will be shared publicly. Audio files will be shared under a data agreement only.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The start date is 2-20-2026. The end date is 50 years later.
Access Criteria: To maximize the benefits of data sharing, the team will share data as broadly as possible to the extent consistent with applicable laws, regulations, rules, and policies. Anyone, including members of the general public, will have access to all of the de-identified data in the form of numbers (e.g., test scores). No video files will be shared. Audio files will be shared with those who qualify and seek permission via a data-sharing agreement. The data-sharing agreement provides for (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. The publicly available data and the data sharing agreement will be accessible in a public-facing Collection in Open Science Framework (osf.io).

REFERENCES:
- Available data/document: Study Protocol — https://doi.org/10.17605/OSF.IO/AJDZS